CLINICAL TRIAL: NCT05470569
Title: Prospective Registry of Patients With Systemic Lupus Erythematosus of the Argentinian Society of Rheumatology
Brief Title: Argentinian Prospective Registry of Patients With Lupus
Status: Recruiting | Type: Observational
Sponsor: Sociedad Argentina de Reumatologia (Other)
Responsible Party: Sponsor
Other Study IDs: RELESSAR PROS
Record Dates: First submitted 2022-07-19; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-06

CONDITIONS: SLE

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Latin America, information about patients with systemic lupus erythematosus (SLE) is limited. Multicenter studies are needed to obtain "real world data '' and to carry out longer follow-ups. The purpose of this project is to design a cohort of Argentinian patients with SLE to describe "our real setting" and to identify possible limitations in access to specialized consultations and treatments.

DETAILED DESCRIPTION:
A longitudinal and multicenter cohort study of patients with systemic lupus erythematosus (SLE) is planned, with a follow-up of for 5 years. The data will be obtained from the clinical history of each patient. The responsible for data collection will always be a physician with experience in the management of patients with SLE and who has received training for data loading.

The data will be collected through the an electronic case report form (eCRF) specially designed for this record and which in turn will facilitate the control of the data and the generation of inquiries to the researchers.

STUDY VARIABLES

Baseline visit:

Sociodemographic data Classification criteria American College of Rheumatology (ACR 1982/1997), Systemic Lupus International Collaborating Clinics (SLICC 2012) and/or European League Against Rheumatism / American College of Rheumatology (EULAR / ACR 2019) History of SLE Access to specialized care Current clinical manifestations Activity and damage Scores Current treatments Patient-Reported Outcomes (PROs): Self-reported quality of life questionnaires EQ-5R; physician global assessment (PGA) and the patient Comorbidities Vaccination Habits Obstetric history Associated antiphospholipid syndrome Hospitalizations for adverse event, infections, or lupus activity

Annual clinical follow-up visits Clinical follow-up of the patient Changes in clinical manifestations Changes in treatments Use of health services; hospitalizations; high cost treatments Activity and damage scores PROs Annual global and SLE-related mortality

STUDY ENDPOINTS

* Number of patients who achieved complete clinical remission or low disease activity status (LDAS)
* Impact on the quality of life and working life measured by PROs and PGA
* Mortality annual and global during the follow up period
* Change in disease activity and damage scores
* Health care resources used reported as number of hospitalizations, emergency visits and need of high cost treatment
* Accessibility to high cost treatment
* Survival of mains drugs reported as time between the first dose and the last dose
* Safety of mains drugs assessed as reason for their discontinuation

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Classified as SLE (according to the 1982/1997 American College of Rheumatology criteria and/or Systemic Lupus International Collaborating Clinics criteria for SLE)
* Less than 5 years from meeting SLE criteria
* Informed consent signature

Exclusion Criteria:

* Diagnosis of other systemic autoimmune diseases or overlap syndromes
* Patients who have been transferred to other centers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with SLE treated and followed up in Rheumatology units belonging to the study group of the Argentine Society of Rheumatology (GESAR-SLE). This is a non-probabilistic sampling study with enrollment of consecutive patients who meet the selection criteria during a one-year enrollment period, added to the patients of RELESSAR I, who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
remission | 1 year
  Number of patients who achieved complete clinical remission or LDAS
patient reported outcomes | 1 year
  Impact on the quality of life and working life measured by PROs
mortality | 1 year
  Annual and global mortality during the follow up period
disease activity | 1 year
  Changes in disease activity (SLEDAI)
accrual damage | 1 year
  change in accrual damage (SLICC)

SECONDARY OUTCOMES:
treatment | 1 year
  Time to high-cost treatment
drug survival | 1 year
  Survival of main drugs reported as time between the first dose and the last dose
adverse events | 1 year
  Safety of main drugs assessed as reason for their discontinuation

CONTACTS AND LOCATIONS:
Locations (1):
- Lucila Garcia, La Plata, Buenos Aires, Argentina